CLINICAL TRIAL: NCT01052285
Title: The Efficacy of Transversus Abdominis Plane Block Versus Placebo Versus Local Infiltration in Patients Undergoing Groin Hernia Repair in Day Case Surgery.
Brief Title: The Efficacy of Transversus Abdominis Plane Block After Groin Hernia Repair
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Glostrup University Hospital, Copenhagen (Other)
Responsible Party: Principal Investigator, Pernille Lykke Petersen, MD, Glostrup University Hospital, Copenhagen
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SM1-plp-10; 2010-018403-29 (EudraCT Number)
Record Dates: First submitted 2010-01-19; First posted 2010-01-20 (Estimated); Last update posted 2011-11-18 (Estimated); Status verified 2011-11

CONDITIONS: Hernia
Keywords: Transversus abdominis plane block
MeSH Terms: conditions — Hernia | interventions — Sodium Chloride; Anesthesia, Local

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo (Placebo Comparator): TAP block with 25 ml of saline Ilioinguinal block with 10 ml of saline and local infiltration with 40 ml of saline.
  Interventions: Procedure: Saline
- Local infiltration (Active Comparator): Ilioinguinal block with 10 ml of ropivacaine 0,375% Local infiltration with 40 ml of ropivacaine 0,375% Tap block with 25 ml of saline
  Interventions: Procedure: Local infiltration
- Transversus abdominis plane block (Experimental): 25 ml of Ropivacaine 0,75%, Ilioinguinal block with 10 ml saline and local infiltration with 40 ml of saline.
  Interventions: Procedure: Transversus abdominis plane block

INTERVENTIONS:
Procedure: Transversus abdominis plane block — UL-guided TAP block with 25 ml of ropivacaine 0,75% unilateral, single dose, ilioinguinal block with 10 ml of saline and local infiltration with 40 ml of saline
  Other Names: postoperative pain, UL-guided block
  Arms: Transversus abdominis plane block
Procedure: Saline — UL-guided Tap block with 25 ml of saline single dose Ilioinguinal block with 10 ml of saline and local infiltration with saline 40 ml single dose
  Other Names: postoperative pain.
  Arms: Placebo
Procedure: Local infiltration — Ilioinguinal block with 10 ml of ropivacaine 0,375% single dose, local infiltration with 40 ml of ropivacaine 0,375% single dose, UL-guided Tap block with 25 ml of saline single dose
  Other Names: Local wound infiltration
  Arms: Local infiltration

SUMMARY:
The purpose of this study is to determine whether Transversus abdominis plane block is superior to placebo or superior to local infiltration in analgesic efficacy after groin hernia repair.

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years old
* groin hernia repair
* written consent
* ASA 1-3
* BMI 18-35

Exclusion Criteria:

* unable to communicate in Danish
* relevant drug allergy
* pain medication in the last 24 hours
* pregnancy
* alcohol or/and drug abuse
* daily opioid intake
* infection at injection site

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2010-06; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Pain scores by coughing between TAP block group and placebo group | 0,2,4,6,8,19 and 24 hours postoperative
  Area under the curve (AUC)-pain during cough based on measurements at 0,2,4,6,8,19,24 hours postoperative

SECONDARY OUTCOMES:
Pain scores by coughing between placebo and local infiltration and between TAP block and local infiltration. | 0,2,4,6,8,19 and 24 hours postoperative
  Area under the curve (AUC)-pain during cough based on measurements 0,2,4,6,8,19,24 hours postoperative.
Total opioid consumption | 0-24 hours postoperative
  Total morphine consumption 0-2 hours postoperative. Total ketobemidone consumption 2-24 hours postoperative.
Postoperative nausea and vomiting | 0,2,4,6,8,19,24 hours postoperative
  Levels of nausea (0-3)at 0,2,4,6,8,19,24 hours postoperative Number of vomits 0-2, 2-4, 4-6, 6-8, 8-19 og 19-24 hours postoperative.
Sedation | 0,2,4,6,8,19,24 hours postoperative
  Levels of sedation (0-3)at 0,2,4,6,8,19,24 hours postoperative.
Pain scores at rest between TAP block versus placebo and TAP block versus infiltration and infiltration versus placebo | 0,2,4,6,8,19,24 hours postoperative
  Area under the curve (AUC)-pain at rest based on measurements at 0,2,4,6,8,19,24 hours postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Pernille L Petersen, MD, Principal Investigator — Glostrup University Hospital
Locations (1):
- Department of Anaesthesiology, Glostrup university hospital, Glostrup Municipality, Denmark

REFERENCES:
- [Derived] Petersen PL, Mathiesen O, Stjernholm P, Kristiansen VB, Torup H, Hansen EG, Mitchell AU, Moeller A, Rosenberg J, Dahl JB. The effect of transversus abdominis plane block or local anaesthetic infiltration in inguinal hernia repair: a randomised clinical trial. Eur J Anaesthesiol. 2013 Jul;30(7):415-21. doi: 10.1097/EJA.0b013e32835fc86f. PMID 23549122